CLINICAL TRIAL: NCT00669955
Title: Efficacy and Safety of Quadruple Therapy by Bismuth Subcitrate Potassium, Metronidazole, and Tetracycline Given X 10 Days With Omeprazole in Eradication of Helicobacter Pylori: A Comparison to Omeprazole, Amoxicillin and Clarithromycin Given X 7 Days
Brief Title: Efficacy and Safety of Quadruple Therapy in Eradication of H. Pylori: A Comparison to Triple Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PYLHp07-01
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2010-08-05 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Helicobacter Infections
Keywords: H. Pylori; Quadruple therapy; Eradication rate; Multinational trial; Resistance to antibiotics; Subjects with confirmed Helicobacter Pylori infection
MeSH Terms: conditions — Helicobacter Infections | interventions — Omeprazole; Amoxicillin; Clarithromycin; Metronidazole; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OAC 7 days (Active Comparator): Triple therapy, given for 7 days at a dose of omeprazole 20 mg twice daily, amoxicillin 500 mg 2 capsules twice daily, and clarithromycin 500 mg 1 tablet twice daily
  Interventions: Drug: Omeprazole, amoxicillin, clarithromycin
- OBMT 10 days (Experimental): OBMT (Pylera), consisting of a 3 in 1 capsule, made of bismuth subcitrate potassium 120 mg, metronidazole 125 mg, and tetracycline 125 mg, administered as 3 capsules 4 times daily. Omeprazole 20 mg is administered twice daily.
  Interventions: Drug: Pylera (Bismuth subcitrate potassium, metronidazole, tetracycline) given in combination with omeprazole

INTERVENTIONS:
Drug: Omeprazole, amoxicillin, clarithromycin — Triple therapy given for 7 days at a dose of omeprazole 20 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID
  Arms: OAC 7 days
Drug: Pylera (Bismuth subcitrate potassium, metronidazole, tetracycline) given in combination with omeprazole — Pylera is a three in one capsule containing bismuth subcitrate potassium 120 mg, metronidazole 125 mg and tetracycline 125 mg given as 3 capsules QID, with omeprazole 20 mg BID.
  Other Names: Pylera
  Arms: OBMT 10 days

SUMMARY:
This study aims at evaluating efficacy and safety of quadruple therapy (bismuth, metronidazole, tetracycline and omeprazole: OBMT) vs triple therapy (amoxicillin, clarithromycin and omeprazole: OAC) in H. Pylori eradication. It is hypothesized that quadruple therapy will be comparable in efficacy to triple therapy. Subjects with confirmed H. pylori positive status will be randomized to one of the treatments described above. At week 6 and 10 follow-up visits, a urea breath test (UBT) will be performed to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 30 days and subjects eligibility will be evaluated after informed consent signature. Endoscopy and Urea Breath test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects assigned to OAC will be treated for 7 days. Those assigned to Pylera will be treated for 10 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 8 and 14.

Follow-up: includes two visits. approximately one and two months post-treatment. Eradication of H. Pylori will be confirmed through UBT, and resistance will be evaluated in case of treatment failure. These subjects will undergo an endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Positive H. Pylori status;
* Presence of upper gastro-intestinal symptoms;
* Mental and legal ability to sign informed consent.

Exclusion Criteria:

* Previous surgery of the GI tract;
* Clinically significant impairment of renal or hepatic function;
* Severe unstable cardiovascular, pulmonary or endocrine disease;
* Barrett's oesophagus or high-grade dysplasia;
* Dysphagia or vomiting as major symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Giguère, PhD, Study Director — Axcan Pharma inc
Locations (1):
- Dr. I. Orpen, Bath, United Kingdom

REFERENCES:
- [Derived] Malfertheiner P, Bazzoli F, Delchier JC, Celinski K, Giguere M, Riviere M, Megraud F; Pylera Study Group. Helicobacter pylori eradication with a capsule containing bismuth subcitrate potassium, metronidazole, and tetracycline given with omeprazole versus clarithromycin-based triple therapy: a randomised, open-label, non-inferiority, phase 3 trial. Lancet. 2011 Mar 12;377(9769):905-13. doi: 10.1016/S0140-6736(11)60020-2. Epub 2011 Feb 21. PMID 21345487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: 11 June 2008 Last patient out: 22 June 2009 Patients were recruited from clinics and hospitals located in seven European Countries: Germany, Poland, Italy, France, Ireland, Spain, United Kingdom.
Pre-assignment Details: If patient was on any contraindicated medications, such as H2 antagonists, sucralfate, or proton pump inhibitors, a washout period of 2 weeks began following informed consent signature, and patient returned to the clinic to perform the endoscopy and the C-13 UBT. Presence of H. pylori needed to be confirmed by C-13 UBT and RUT at least.
Groups:
- Quadruple Therapy (OBMT) 10 Days: Omeprazole 20 mg BID (twice a day), and the 3 in 1 capsule, Pylera, containing Bismuth Subcitrate potassium 140 mg, metronidazole 125 mg and tetracycline 125 mg, administered as 3 capsules QID (four times day)
- Triple Therapy (OAC) 7 Days: Omeprazole 20 mg BID, Amoxicillin 500 mg 2 capsules BID and Clarithromycin 500 mg 1 tablet BID
Period: Overall Study
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Started | 218 (216 patients received study drug. 2 patients were dispensed study drug but did not take it) | 222
Completed | 204 | 195
Not Completed | 14 | 27
Not completed — Adverse Event | 3 | 5
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 5 | 7
Not completed — Protocol Violation | 2 | 7
Not completed — Investigator Sponsor Judgement | 0 | 1
Not completed — not compliant with study drug/visit | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days | Total
Number analyzed (Participants) | 218 | 222 | 440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 184 | 194 | 378
  >=65 years | 34 | 28 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.53 (14.64) | 47.95 (14.52) | 48.24 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 100 | 205
  Male | 113 | 122 | 235
Region of Enrollment [Number; unit: participants]
  Italy | 10 | 10 | 20
  Spain | 7 | 6 | 13
  France | 15 | 17 | 32
  Germany | 92 | 91 | 183
  Poland | 91 | 93 | 184
  United Kingdom | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Helicobacter Pylori Eradication Confirmed by Urea Breath Test
Description: H. pylori Eradication defined as a negative C13-UBT (urea breath test) result at both Week 6 and Week 10 follow-up visits.
Time Frame: Week 6 and week 10 follow-up visits
Population: No imputation method used, as this is the per protocol population, which excludes patients with missing values, or with protocol violations.
Measure: Number; unit: Participants
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Number analyzed (Participants) | 178 | 161
Participants | 166 | 112

2. Secondary Outcome: Number of Patients Experiencing Treatment Emergent Adverse Events.
Description: A treatment-emergent adverse event is defined as an event not present prior to exposure to the study medication or any event already present that worsens in either intensity or frequency following exposure to study medication up to 30 days after study discontinuation.
  All safety analysis based on the safety population.
Time Frame: at the end of treatment (day 8-14), week 6 and wek 10 follow-up visits.
Population: Safety population, described as all randomized patients having received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Number analyzed (Participants) | 216 | 222
Participants | 101 | 112

3. Secondary Outcome: H. Pylori Eradication and Presence or Past History of Peptic Ulcers
Description: Eradication rates in the subset of patients with peptic ulcer (current or past history) at baseline are reported based on the per protocol population. Eradication must be confirmed at week 6 and week 10 by a negative Urea Breath Test conducted within the allocated windows.
Time Frame: Week 6 and week 10 follow-up visits
Population: Per protocol population.
Measure: Number; unit: Participants
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Number analyzed (Participants) | 19 | 18
Participants | 18 | 15

4. Secondary Outcome: Clarithromycin Resistance
Description: Eradication rates in subset of patients infected with a bacterial strain confirmed as resistant to clarithromycin at baseline. Resistance to clarithromycin defined as Minimum Inhibitory Concentration (MIC) of 1 ug/ml and above
Time Frame: Measured at baseline
Population: Per protocol analysis population
Measure: Number; unit: participants
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Number analyzed (Participants) | 33 | 25
participants | 30 | 2

5. Secondary Outcome: Metronidazole Resistance
Description: Eradication rates in subset of patients infected with a bacterial strain confirmed as resistant to metronidazole at baseline. Resistance to metronidazole defined as Minimum Inhibitory Concentration (MIC) above 8 ug/ml
Time Frame: Measured at baseline
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Number analyzed (Participants) | 42 | 41
participants | 38 | 28

6. Secondary Outcome: Overall Compliance to Study Medications
Description: Overall compliance: number of capsules dispensed - number of capsules returned/Number of prescribed capsules X 100. Percentages based on safety population
Time Frame: At the end of the treatment phase (days 8-14)
Population: Safety population.
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Number analyzed (Participants) | 216 | 218
participants | 97.58 (10.71) | 97.47 (14.91)

7. Secondary Outcome: Number of Patients With Bismuth Plasma Concentrations Above the Toxic Level
Description: Tolerability of OBMT with respect to plasma bismuth concentrations: number of patients with bismuth concentrations above the toxic level (50 ug per liter)
Time Frame: Baseline (both arms), end of treatment (Day 11-14) and end of study (Day 70) OBMT arm only
Population: Plasma bismuth concentrations were analysed in the OBMT arm only. The goal was to determine whether bismuth plasma concentrations would be of 50 ug/l or above at end of treatment, or at the end of study. The results report the number of patients having reached 50 ug/l in the OBMT arm at either of these timepoints.
Measure: Number; unit: participants
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Number analyzed (Participants) | 216 | 0
participants | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events were recorded starting at the signing of the informed consent until the final visit (Day 70) or early withdrawal visit. Serious adverse events were followed until 30 days after the patient had stopped study participation.
Description: Systematic assessment done for laboratory evaluations and bismuth plasma levels.
Arm/Group | Quadruple Therapy (OBMT) 10 Days | Triple Therapy (OAC) 7 Days
Serious Adverse Events (participants affected / at risk) | 4/216 | 3/222
Other Adverse Events (participants affected / at risk) | 98/216 | 105/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadruple Therapy (OBMT) 10 Days (N=216) | Triple Therapy (OAC) 7 Days (N=222)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
e coli urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quadruple Therapy (OBMT) 10 Days (N=216) | Triple Therapy (OAC) 7 Days (N=222)
Dyspepsia (Gastrointestinal disorders) | 22 | 30
Diarrhea (Gastrointestinal disorders) | 14 | 28
Abdominal pain upper (Vascular disorders) | 18 | 16
Nausea (Gastrointestinal disorders) | 14 | 2
Dysgeusia (Nervous system disorders) | 12 | 22
Headache (Gastrointestinal disorders) | 18 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with the agreement with investigators. Axcan will allow publication after a multi-centre publication or after an agreed period, subject to review by Axcan for confidentiality and intellectual protection.